CLINICAL TRIAL: NCT00545207
Title: A Randomized, Double-blind Study of the Effect of Oral Monthly Bonviva on in Vivo Bone Micro-architecture Parameters in Post-menopausal Women With Osteopenia
Brief Title: A Study of Bonviva (Ibandronate) Once Monthly in Post-Menopausal Women With Osteopenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML19357
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Post-Menopausal Osteopenia
MeSH Terms: interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 2 years
  Arms: 1
Drug: Placebo — po monthly for 2 years
  Arms: 2

SUMMARY:
This 2 arm study will compare the effect of oral Bonviva (150mg, monthly) and placebo on parameters of bone micro-architecture, assessed by CT scan, bone turnover and bone mineral density. Patients will be randomized to receive either Bonviva 150mg po or placebo monthly, and measurements will be taken at baseline, and at intervals over 2 years. The anticipated time on study treatment is 2+ years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women, aged 55-75 years;
* diagnosed osteopenia.

Exclusion Criteria:

* history of osteoporotic vertebral fracture;
* contraindication to ibandronate.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Trabecular BV/TV at distal radius of non-dominant arm | 12 arms

SECONDARY OUTCOMES:
Trabecular BV/TV at distal radius of non-dominant arm | 6 months and 2 years
Bone density, trabecular BV/TV at distal tibia | 6 months, 1 and 2 years
Serum CTX | Intervals throughout study
Lumbar hip and wrist BMD | 1 and 2 years
AEs and laboratory parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- France (4):
  - Lyon
  - Paris
  - Saint-Priest-en-Jarez
  - Toulouse